CLINICAL TRIAL: NCT00402974
Title: The VITAKIDS-Study: The Effect of Vitamin K Supplementation on Osteocalcin Carboxylation in Healthy Children
Brief Title: The Effect of Vitamin K Supplementation on Osteocalcin Carboxylation in Healthy Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL14210.000.06; METC Utrecht: 06/232
Record Dates: First submitted 2006-11-21; First posted 2006-11-23 (Estimated); Last update posted 2008-06-10 (Estimated); Status verified 2008-06

CONDITIONS: Healthy
Keywords: osteocalcin; vitamin K; carboxylation; healthy children
MeSH Terms: interventions — menaquinone 7

INTERVENTIONS:
Drug: menaquinone 7

SUMMARY:
Background of the study:

Results from several studies show that vitamin K has an important function in bone metabolism. In a previous cross-sectional study conducted by our department, evidence for a poor vitamin K status of bone during growth in children was found (unpublished data, accepted for publication Pediatric Research, october 2006). These findings justify clinical intervention studies in which bone quality is monitored as a function of long-term vitamin K-supplementation. Before a long-term intervention study is undertaken, it is important to determine the effect of vitamin K administration on osteocalcin carboxylation in this specific population. Although the relationship between increased vitamin K intake and osteocalcin carboxylation was already clearly demonstrated in several adult groups (e.g. healthy adults, postmenopausal women), this has never been shown in children.

Objective of the study:

To study the effect of a vitamin K-containing food supplement (menaquinone 7) on osteocalcin carboxylation in healthy children between 6 and 10 years of age in the Netherlands.

Study design:

Randomised double-blind placebo-controlled intervention study.

Study population:

55 healthy children (boys and girls) between 6 and 10 years, recruited from primary schools.

Intervention:

The subjects are randomised into two groups:

* placebo group: during 8 weeks, 27 children will receive one tablet of placebo- food supplement per day
* treatment group: during 8 weeks, 28 children will receive one tablet of food supplement per day containing 45 µg vitamin K2.

Primary study parameters/outcome of the study:

Undercarboxylated (ucOC) and carboxylated (cOC) fractions of osteocalcin will be measured by enzyme-linked immunosorbent assay (ELISA). Both the ucOC fraction and the ucOC/cOC ratio (UCR) are sensitive indicators for the vitamin K status of bone. Elevated levels of UCR are indicative of an inferior vitamin K status of bone. The main study parameters are the mean percentages of change in serum undercarboxylated osteocalcin (ucOC) and UCR from baseline (t=0) to endpoint (t=8 weeks) in both treatment groups.

Secondary study parameters/outcome of the study (if applicable):

The secondary end points are the percentages of change in serum vitamin K levels in relation to lipid metabolism markers from baseline to endpoint in each individual.

Furthermore, the percentages of changes in serum BAP and NTX from baseline to endpoint in each individual are considered to be endpoints as well.

ELIGIBILITY:
Inclusion Criteria:

* Healthy prepubertal male and female children
* Subjects of normal body weight and height according to standard Dutch growth charts (within p3-p97)
* Subject and/or parent of subject has given written consent to take part in the study

Exclusion Criteria:

* Subjects with (a history of) metabolic or gastrointestinal disease
* Subjects with (a history of) soy allergy
* Subjects using vitamin supplements containing vitamin K
* Subjects presenting chronic inflammatory diseases
* Subjects receiving systemic treatment or topical treatment likely to interfere with evaluation of the study parameters
* Subjects receiving corticoϊd treatment
* Subjects using oral anticoagulants

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2007-01; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
mean percentages of change in serum undercarboxylated osteocalcin (ucOC) and UCR from baseline (t=0) to endpoint (t=8 weeks) in both treatment groups

SECONDARY OUTCOMES:
percentages of change in serum vitamin K levels in relation to lipid metabolism markers from baseline to endpoint in each individual
the percentages of changes in serum BAP and NTX from baseline to endpoint in each individual

CONTACTS AND LOCATIONS:
Overall Officials: Wietse Kuis, PhD MD, Principal Investigator — WKZ, UMC Utrecht
Locations (1):
- Wilhelmina Children's Hospital (WKZ), University Medical Center (UMC) Utrecht, Utrecht, Netherlands